CLINICAL TRIAL: NCT06163313
Title: Retrospective and Prospective Study of Patients Suffering From Nephrolithiasis Undergoing Surgery Using a Minimally Invasive Endoscopic Approach.
Brief Title: Protocol No. 2016 - Calculosis- Endourology;
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Professor, IRCCS San Raffaele
Other Study IDs: 2016 - Calcolosi
Record Dates: First submitted 2023-11-21; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Calculosis
Keywords: calculosis; calculi; endourologia
MeSH Terms: conditions — Lithiasis; Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Calculosis patients: Patients suffering from kidney stones
  Interventions: Other: Observation of patients suffering from kidney stones who undergo endoscopic surgery

INTERVENTIONS:
Other: Observation of patients suffering from kidney stones who undergo endoscopic surgery — Clinical data will therefore be acquired through a collection of medical history, physical examination, blood chemistry and instrumental test reports;

SUMMARY:
Retrospective and prospective study on patients suffering from nephrolithiasis who undergo minimally invasive surgery of the upper excretory system; correlation between the phenotypic and genotypic aspects of the patients and the stone pathology treated with an endoscopic surgical approach.

DETAILED DESCRIPTION:
Clinical data will be collected from patients suffering from kidney stones before and after surgery, in order to demonstrate how the endoscopic approach can not only be effective in treating kidney stones but also reduce operative complications.

These data will be collected in a database in order to be able to perform statistical analyzes useful for demonstrating our theory.

Furthermore, data from the surgery will be collected regarding the endoscopic instruments used and the intraoperative findings (site, size, appearance of the stone), degree of calcification of the renal papillae.

All this in order to improve the therapeutic approach to patients suffering from stones and reduce the risk of recurrence over time through the identification of genetic expression patterns that predispose to the expression of the stone phenotype.

ELIGIBILITY:
Inclusion Criteria:

* subjects suffering from kidney stones or tumors of the upper excretory tract >= 18 years
* signature of informed consent

Exclusion Criteria:

* subjects < 18 years
* presence of mental or physical disability that may prevent the patient from answering the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from kidney stones who undergo endoscopic surgery
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2016-09-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2066-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical data | Baseline and after 6 months
  Medical history: patient's medical history, past surgical history, family medical history, social history, allergies, and medications; physical examination: vital signs, temperature examination, blood pressure, pulse, and respiratory rate blood chemistry and instrumental test reports: Serum PSA levels, conventional imaging
Eating habits | Baseline and after 6 months
  Eating habits through an ad-hoc eating habits questionnaire
Prostatic Function | Baseline and after 6 months
  Prostatic Function through the International Prostatic Symptoms Score questionnaire, IPSS, Scoring 0 -7, 0-7 mild symptoms, 8-19 moderate symptoms, 20-35 severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Salonia, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No